CLINICAL TRIAL: NCT02789761
Title: The Vascular and Cognitive Effects of Chronic High-flavanol Intake in Healthy Males
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor of Biochemistry, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MCStudy
Record Dates: First submitted 2016-04-25; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: Flow-mediated dilatation (FMD); Vascular function; cognitive function

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-flavanol milk chocolate (Active Comparator): Bi-daily consumption of 12 g portion of a high-flavanol milk chocolate containing approximately 35 mg of (-)-epicatechin for 2-weeks (14 days)
  Interventions: Dietary Supplement: High-flavanol milk choocolate
- Low-flavanol milk chocolate (Placebo Comparator): Bi-daily consumption of 12 g portion of a low-flavanol milk chocolate containing approximately <1 mg of (-)-epicatechin for 2-weeks (14 days)
  Interventions: Dietary Supplement: Low-flavanol milk chocolate

INTERVENTIONS:
Dietary Supplement: High-flavanol milk choocolate
  Other Names: Epicatechin-rich milk chocolate
  Arms: High-flavanol milk chocolate
Dietary Supplement: Low-flavanol milk chocolate
  Arms: Low-flavanol milk chocolate

SUMMARY:
A randomised, placebo-controlled, parallel human dietary intervention trial conducted in 33 healthy males to investigate the vascular and cognitive effects of bi-daily consumption of high-flavanol (epicatechin-rich) milk chocolate over a 2-week intervention period. Subjects visited the Hugh Sinclair Unit of Human Nutrition on 3 separate occasions; at the beginning, end and post-intervention.

ELIGIBILITY:
Inclusion Criteria

* Body Mass Index 18.5-27.5 kg/m2
* Normal Blood pressure (< 150/90)
* Non-smoker
* Regular exercise routine
* Signed consent form

Exclusion Criteria:

* Haemoglobin (anaemia marker) < 125 g/l
* Gamma GT (liver enzymes) > 80 IU/l
* Total Cholesterol > 6.5 mmol/l
* Suffered a myocardial infarction or stroke in the last 12 months
* Suffers from any cardiovascular or metabolic disorders
* Suffers from any blood-clotting disorder, and/or takes supporting medication
* Any dietary restrictions or on a weight reducing diet
* On any lipid-modifying or blood pressure lowering medication
* Consuming any specific vitamin/ herbal supplements or fish oils

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Flow-mediated Dilation (FMD) | Change from baseline at 14 days
  Ultrasound-based assessment of brachial artery reactivity following induced reactive hyperemia

SECONDARY OUTCOMES:
Blood pressure (BP) | Change from baseline at 14 days
  Acute assessment of systolic and diastolic BP (3 repeats)
Executive Function | Change from baseline at 14 days
  Assessed by cognitive test battery
Endothelial progenitor cells and Microparticles | Change from baseline at 14 days
  Flow cytometric analysis using whole blood
Plasma flavanol metabolite analysis | Change from baseline at 14 days
  HPLC-MS assessment of metabolite profile and content of plasma
Plasma Nitrite & Nitrate analysis | Change from baseline at 14 days
  HPLC-based system with inbuilt colorimetric Griess reaction assay for the assessment of Nitrite & Nitrate in plasma
Serum analysis of cardivascular-related blood marker(s) concentration | Change from baseline at 14 days
  ILAB assessment of serum content of glucose, Triglycerides, total cholesterol, HDL-cholesterol, C-reactive protein and Non-esterified fatty acids
Serum analysis of insulin | Change from baseline at 14 days
  ELIZA kits for determination of insulin concentration in serum

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy P Spencer, PhD, Principal Investigator — Univerisity of Reading

IPD SHARING:
Plan to Share IPD: No